CLINICAL TRIAL: NCT02489825
Title: Pilot Study: Does Preventive Adjacent Level Cement Augmentation Positively Affect Reoperation Rates After Osteoporotic Vertebral Compression Fractures?
Brief Title: Study About the Effect of Preventive Adjacent Level Cement Augmentation After Osteoporotic Vertebral Compression Fractures
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Death of study initiator
Sponsor: University of Bern (Other)
Collaborators: Sonnenhof Hospital, Bern (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 008/13; 13-01-F (Other Grant/Funding Number: Lindenhofstiftung Bern)
Record Dates: First submitted 2015-06-25; First posted 2015-07-03 (Estimated); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Osteoporosis; Vertebral Fracture
Keywords: randomized controlled trial; vertebral fracture; osteoporosis; vertebroplasty; augmentation
MeSH Terms: conditions — Osteoporosis; Spinal Fractures

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Augmentation vertebroplasty (Other): Single level fracture fixation with vertebroplasty
  Interventions: Procedure: Augmentation vertebroplasty
- Augmentation and prophylactic vertebroplasty (Other): Triple level augmentation with VP fixation of the fracture and additional prophylactic vertebroplasty in both the adjacent levels
  Interventions: Procedure: Augmentation and prophylactic vertebroplasty

INTERVENTIONS:
Procedure: Augmentation vertebroplasty — Cement augmentation of fractured vertebral body
  Arms: Augmentation vertebroplasty
Procedure: Augmentation and prophylactic vertebroplasty — Cement augmentation of fractured vertebral body and prophylactic augmentation of both adjacent vertebral bodies
  Arms: Augmentation and prophylactic vertebroplasty

SUMMARY:
Vertebroplasty itself is challenged regarding its clinical efficacy. While two randomized controlled trials (RCTs) with substantial methodological problems have led to an intense discussion another RCT with larger case numbers, more representative inclusion criteria and a more consistent and sound methodology has revealed results that mirror the investigators' own clinical experience. In their daily practice, the investigators have further advanced their treatment concept and routinely apply prophylactic augmentations with VP using an algorithm. Biomechanical studies support their approach, but clinical studies are rare so far. Prophylactic augmentation with balloon kyphoplasty has not shown convincing effects in a small pilot study. Given the above mentioned methodological and clinical disputes and the call for high-evidence studies about VP, the investigators aim at generating a reliable sample size calculation and preliminary results for a future multicenter RCT about prophylactic adjacent level augmentation with VP in single level osteoporotic compression fractures.

DETAILED DESCRIPTION:
Background

Despite current academic debates percutaneous vertebroplasty (VP) has been convincingly used for the treatment of osteoporotic compression fractures all around the world. Polymethylmethacrylate bone cement is directly injected into a fractured vertebral body through one or two bone biopsy needles to stabilize the fracture fragments and to possibly improve the vertebral body height. The fracture pain represents a significant burden for the patients, limiting physical function, quality of life and increasing social isolation.

The immediate and clinically relevant pain alleviation after vertebroplasty does therefore have a large impact on patients' mobility, autonomy and quality of life.

The current state of the art in the treatment of acute osteoporotic vertebral compression fractures that are nonresponsive to conservative treatment is still augmentation of the fractures with VP or balloon kyphoplasty (BKP) given an intact posterior vertebral body wall. BKP is claimed to be saver by reducing the occurrence of cement leakages and more effective in reducing the fracture, i.e. reconstituting vertebral body height. While the first argument largely depends on the definition of an adverse event, i.e. is an asymptomatic radiologically visible cement leakage truly a complication, the second argument could not hold its promise since the regained vertebral body height is partially lost after balloon deflation. This problem is tackled by further developed BKP technologies like vertebral body stenting (VBS). From a cost-effectiveness perspective, VP is superior to conservative medical care and one can postulate that it is hence also more cost-effective than BKP which is a much more costly treatment option.In addition, it is the only prophylactic augmentation option that does not "destroy" intact unfractured bone structures by deployment of the balloon but does only augment them. It is hence the least aggressive augmentation option for prophylaxis.

Osteoporosis as the underlying disease leads to an increased risk of fractures of the adjacent vertebral bodies, with incidences up to 22% in the first year. After fracture augmentation new fractures in the spine can occur. This leads to reoperations in a frail population with high numbers of American Society of Anaesthesiologists (ASA) 3-4 patients. Any non-life-saving surgical intervention in these patients needs to be avoided. Therefore, prophylactic augmentation of the adjacent non-fractured vertebral bodies is a treatment option which is safe and may reduce reoperation rates. Since VP is currently under scientific and clinical scrutiny and calls for level-one-evidence become audible everywhere, the investigators plan to assess the hypothesis that prophylactic augmentation significantly decreases reoperation rates for adjacent new fractures with a randomized controlled trial.

Objective

The aim of the proposed study is to show the effect of preventive augmentations of adjacent vertebral bodies on 6 (12) months reoperation rates.

Subjects with an acute (<= 6 weeks) single level osteoporotic compression fracture, meeting the inclusion criteria and having no exclusion criterion will be randomized to either single level fracture fixation with vertebroplasty or triple level augmentation with VP fixation of the fracture and additional prophylactic vertebroplasty in both adjacent levels. The hypothesis is that prophylactic VP augmentation of both adjacent vertebral bodies in acute single level osteoporotic compression fractures results in significantly lower reoperation rates for new spinal fractures within 6 months after surgery compared to isolated single level fracture fixation.

Methods

This is an open label mono-center randomized controlled pilot trial. Given the timeframe and budget of the study, the investigators aim at conducting a pilot trial for clinically verifying the sample size calculation in order to have a sound basis of information for planning a larger multicenter trial. The inclusion of primary cases will last for 12 months, the followup intervals for each case will be 2 and 6 months since the large majority of new fractures appears within that time window. 12 months followup will be conducted by mail/telephone interview. Preliminary calculation of results, i.e. a new corrected sample size will hence be carried out at the end of one and a half years. Two treatment groups will be compared:

Group 1: single level fracture fixation with vertebroplasty, Group 2: triple level augmentation with VP fixation of the fracture and additional prophylactic vertebroplasty in both the adjacent levels.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 55 years
* Written informed consent
* Single level acute (< 6 weeks) vertebral compression fracture
* Fracture due to diagnosed or presumed underlying primary or secondary osteoporosis
* Patients with Association for the study of Osteosynthesis (AO) type A1.x fractures and A3.1 fractures may be included in the study
* Target Vertebral Compression Fracture (VCF) is between T10 and L4
* Target VCF to be treated shows either: height change - an acute (< 6 weeks) change in VB height (>15% height loss) with height loss at the anterior or middle portion of the VB consistent with a worsening of 1 or more grades acc to Genant
* OR positive MRI or bone scan - VB shows hyperintense signal on MRI-T2 or STIR sequence
* OR target VB is positive on radionuclide bone scan
* Back pain correlating with the location of the VCF
* Treatment of target and adjacent VCFs is technically feasible by and clinically appropriate for vertebroplasty
* No previous VCFs
* No major surgery of the spine planned for at least 6 months following enrollment
* Pre-treatment back pain by numerical rating scale (NRS) score > 4 (0-10 scale)
* Subject is able to understand the risks and benefits of participating in the study and is willing to provide written informed consent
* Psychosocially, mentally and physically able to fully comply with the protocol requirements for the duration of the study including adhering to scheduled visits, treatment plan, completing forms and other study procedures.

Exclusion Criteria

* VB morphology or configuration is such that vertebroplasty is not technically feasible for the targeted and adjacent VCFs
* Fracture due to high-energy trauma
* Suspected OR proven cancer inside index vertebral body
* Disabling back pain due to causes other than acute fracture (e.g., sacroiliac fracture, symptomatic degenerative disc disease, lumbar spinal stenosis)
* Any painful VCF with fracture age > 6 weeks
* Patients with primary tumors of the bone (e.g., osteosarcoma) or solitary plasmacytoma at site of the index or adjacent VCF
* Any objective evidence of neurologic compromise at baseline.
* Previous balloon kyphoplasty, VBS or vertebroplasty for any VCF
* Significant clinical comorbidity that may potentially interfere with follow-up (e.g., dementia, severe comorbid illness)
* Patients requiring the use of high-dose steroid (>= 100mg prednisone or 20 mg dexamethasone per day), IV pain medication, or nerve block to control chronic back pain unrelated to index VCF
* Spinal cord compression or canal compromise requiring decompression
* Patients with osteoblastic tumors at the site of the index VCF
* MRI contraindication (e.g. cerebral aneurysm clips, pacemaker, implanted biostimulators, cochlear implants, penile prosthesis)
* Spinal instability as indicated by neurologic deficit, kyphosis >30°, compression >50%, translation >4 mm, interspinous-process widening.
* Pre-existing conditions contrary to vertebroplasty, such as: irreversible coagulopathy or bleeding disorder
* Allergy to bone cement.
* Any evidence of VB or systemic infection

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2022-02 (Actual); Study Completion 2022-02 (Actual)

PRIMARY OUTCOMES:
Number of new operations within 6 months after vertebroplasty due to adjacent or distant segment fracture. | 6 months after index surgery
  Measured by interview, clinical & radiographic assessment

SECONDARY OUTCOMES:
Disease specific quality of life (COMI back form) | 6 months after index surgery
  Measured by questionnaire
General quality of life | 6 months after index surgery
  Measured by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Paul Heini, MD, professor, head of dept., Principal Investigator — Sonnenhof Hospital, Bern
Locations (1):
- Sonnenhof hospital, dept. of spinal surgery, Bern, Switzerland

REFERENCES:
- [Result] Diel P, Freiburghaus L, Roder C, Benneker LM, Popp A, Perler G, Heini PF. Safety, effectiveness and predictors for early reoperation in therapeutic and prophylactic vertebroplasty: short-term results of a prospective case series of patients with osteoporotic vertebral fractures. Eur Spine J. 2012 Aug;21 Suppl 6(Suppl 6):S792-9. doi: 10.1007/s00586-011-1989-x. Epub 2011 Aug 30. PMID 21877131